CLINICAL TRIAL: NCT05982184
Title: Effect of Music Prehabilitation on Preoperative Anxiety in Patients Undergoing Colorectal Oncological Resection: a Multicentre Randomized Controlled Trial
Brief Title: Effect of Music Prehabilitation on Preoperative Anxiety Before Surgery
Acronym: MU-PRIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Markus Klimek, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9411
Record Dates: First submitted 2023-07-14; First posted 2023-08-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cancer of Colon; Surgery; Anxiety
Keywords: Music; Colon cancer; Surgery; Anxiety; Perioperative care; Prehabilitation; Non pharmacological intervention
MeSH Terms: conditions — Colonic Neoplasms; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Music intervention at home. Patients will be asked to listen to music using their own equipment three times a day. Starting approximately a week prior to surgery up to the day of surgery.
  Interventions: Other: Music
- Standard Care (No Intervention): Treatment as usual.

INTERVENTIONS:
Other: Music — Patient preferred music listened to through earpieces or headphones using patients' own hardware and software.
  Other Names: Music medicine; music intervention
  Arms: Music

SUMMARY:
The goal of this multicenter randomized controlled trial is to investigate the effect of music prehabilitation on preoperative anxiety in patients undergoing elective oncological colorectal resection. Patients will be asked to listen to music three times a day starting one week before day of surgery. Anxiety levels will be compared with the control group that is not explicitly instructed to listen to music by using validated questionnaires

DETAILED DESCRIPTION:
Perioperative music interventions have been proven to have a positive effect on surgical patients regarding postoperative pain, anxiety and stress. Preoperative anxiety is a predictor for postoperative pain. It is hypothesized that preoperative anxiety develops at home. Unfortunately, data on this subject is scarce. Prehabilitation is a relatively new concept, which improves the patient's condition at home waiting for a surgical intervention. No studies exist in which music is implemented as a prehabilitation method. Music interventions are relatively simple low cost, sustainable and know no side effects. The researchers hypothesize that the use of pre-admittance music interventions as a prehabilitation modality in oncological colorectal surgical patients will decrease preoperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 16 years
* Patients undergoing elective oncological colorectal surgery at participating center
* Minimal hospital stay of 2 days postoperatively.
* Sufficient knowledge of the Dutch language
* Communicable and able to assess the questionnaires
* Patients who have access to personal music playing device and headphones/earphones. - Written informed consent acquired from the patient

Exclusion Criteria:

* Patients with severe hearing impairment (defined as no or barely verbal communication possible).
* Patients with an expected stay of less than two nights in the hospital
* Patients who are professional musicians.
* Active music players or singers who may play or sing every week
* Patients who actively listen to music with a duration of > 30 minutes daily. Active listening is defined as music listening with headphones/earphones, while this is not combined with any other activity (e.g. exercising, working, driving or religious activities).
* Patients who have a preoperative waiting period of less than five days.
* Participation in another study that may possibly intervene with the outcome measures. (e.g. use of psychiatric medication during inclusion or prehabilitation interventions or similar procedures according to the judgement of the research team)
* Assessment of primary outcome is not possible.
* Patients with mental disorders influencing their ability to adhere to the study protocol and/or assess the questionnaires.
* Inability or unwillingness to receive the music intervention.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-11-22 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Patient reported anxiety measured by the 6-item Spielberger State-trait Anxiety (STAI-6) inventory at admission. | Baseline and day of admittance to hospital
  The STAI-6 questionnaire is a validated and frequently used six item questionnaire to assess anxiety. Six questions regarding feelings of anxiety are scored on a four point Likert scale. Scoring is achieved by reverse scoring of the positive items, sum all six scores, and multiplying the score by 20 divided by 6. The score ranges between 20 and 80, in which a higher score correlates with a higher anxiety level.

SECONDARY OUTCOMES:
Patient reported pain on a 1-10 numeric scale. | Thrice daily on each post-operative day until discharge
  Pain scores are gathered thrice daily by nurses as part of standard care
Incidence of delirium diagnosis made by geriatricians or psychiatrists | Post-operative until discharge
  Diagnosis of delirium by geriatricians or psychiatrists as noted in the electronic health report were considered as a confirmed diagnosis of delirium
Delirium observation scale scores (DOS). | Post-operative until discharge
  The DOS is a 13-point screen for delirium, based on Diagnostic and statistical manual of mental disorders version 4 (DSM-IV) delirium criteria, designed to be completed by a nurse. Responses are dichotomous. Scores ≥ 3 were considered positive delirium screens.
Subjective stress, measured with the 10-item perceived stress scale (PSS-10) questionnaire at baseline, day of admittance and at discharge. | Baseline, day of admittance and discharge
  The PSS-10 is a validated questionnaire which assess subjective stress. It is a 10-item, comprehensive, reliable and valid instrument which is created and validated in the American population and widely used in medical/psychological studies. The items are each scored on a five-point Likert scale (ranging from 0 = never to 4 = very often). A Dutch translation of the PSS-10 was created according to the principles of good translation (the existing English version was translated to Dutch by a native Dutch speaker, afterwards the translated Dutch version was compared to the original validated English version by a native English speaker)(
Quality of life at 30 days postoperatively, measured with the EuroQol-5dimension-5length EQ-5D-5L questionnaire. | 30 days postoperatively
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The descriptive system comprises five dimensions. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Rate, timing and total dosages of medication given to the patient (sedatives, analgetics etc.) | From admission to discharge
  Every medication and dose provided to the patient is recorded in the EHR and will be extracted to assess possible differences in medication requirements between intervention and control group
A self-made questionnaire assessing patient satisfaction regarding music intervention | 4 weeks postoperatively at follow-up
  A 5-item questionnaire comprised of dichotomous and open ended questions regarding the patients satisfaction with the music intervention.
Rate of complications | Postoperatively until 30 days follow-up
  Complication documentation as provided my medical staff and associated Clavien-Dindo score
Quality of recovery is a comprehensive 40-item questionnaire (QoR-40) used to assess the rate of recovery after surgery. | 4 weeks postoperatively at follow-up
  The quality of recovery will be assessed using de QoR-40 questionnaire, assessed at 30 days postoperatively. This is a questionnaire which assesses five subscales, including emotional state, physical independence, psychological support, pain and physical comfort. The questionnaire uses a five-point Likert scale.

OTHER OUTCOMES:
Age | At moment of surgery
  In years
Sex | at baseline
  Male/Female
BMI | At admittance
  Quetelet index
Surgery characteristics | Intraoperatively
  Duration, type of procedure.
Prior medical history | At baseline
  Previous diagnoses, treatment
Music preferences in daily life. An 8-item researcher made questionnaire. | At baseline
  Items explore music listening activities, preferences for musical genres and potential music playing background. Question types varies from dichotomous answers to radio buttons, and dropdown lists.
Length of sedation in minutes | Perioperatively
  Length of peroperative sedation as recorded in EHR by attending anesthesist
Rate and type of complications during surgery as recorded in the EHR | From entering the operation room to exit to postoperative nursing ward of post-anesthesia care unit (PACU)
  Complications that occur during the surgery are recorded in the EHR and will be extracted

CONTACTS AND LOCATIONS:
Overall Officials: Markus Klimek, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- Netherlands (5):
  - Amphia Ziekenhuis, Breda, North Brabant
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Franciscus Gasthuis, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Admiraal de Ruyter Ziekenhuis, Goes, Zeeland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verhoeven JG, Geensen R, Dirven TLA, Rietdijk WJR, Birnie E, Jeekel J, Klimek M. Study protocol for a multicentre randomised controlled trial using music prehabilitation to reduce preoperative anxiety before oncological colorectal surgery: the MU-PRIOR trial. BMJ Open. 2025 Apr 29;15(4):e095239. doi: 10.1136/bmjopen-2024-095239. PMID 40306915